CLINICAL TRIAL: NCT04226937
Title: DLBCL Interim Response Evaluation for Customised Therapy
Acronym: DIRECT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Collaborators: AstraZeneca (Industry); Cancer Research UK Cambridge Institute (Other)
Responsible Party: Principal Investigator, Daniel Hodson, Dr, Cambridge University Hospitals NHS Foundation Trust
Other Study IDs: DIRECT
Record Dates: First submitted 2020-01-06; First posted 2020-01-13 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: High-grade B-cell Lymphoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — ctDNA and Biopsy Tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Not Applicable as this is a translational, sample collection study. — Patients will take their normal standard of care treatment for their lymphoma, as per agreed with the patient's doctor.
  Blood samples will be collected at Baseline, during the first 3 cycles of Treatment, at End of Treatment, at 6- and 12-months after End of Treatment and at relapse/progression if applicable.
  Surplus Tissue biopsy will be collected at Baseline and at relapse/progression if applicable. In rare cases research-specific tissue biopsy may be collected if appropriate.

SUMMARY:
The aim of the DIRECT Study is to establish a robust pipeline to identify those patients with high-grade B cell lymphoma most suitable for novel agent clinical trials based upon genomic subtype and an integrated response evaluation determined early in first-line therapy.

DETAILED DESCRIPTION:
This will be done by integrating data and samples collected from patients undergoing standard of care treatment for high-grade B cell lymphoma

Data will be integrated from

1. Clinical risk factors from the International Prognostic Index (IPI)
2. Up-front genomic subtype based on molecular profiling of diagnostic biopsy
3. Serial ctDNA monitoring during treatment.
4. Radiological response imaging

ELIGIBILITY:
* Have given written informed consent to participate.
* Age ≥ 18 years at the time of consent.
* Histologically confirmed diagnosis of previously untreated high-grade B cell lymphoma.
* Planned to receive immunochemotherapy as first-line therapy, e.g. R-CHOP therapy.
* Planned or completed standard of care imaging (CT or PET-CT)
* Able to give blood.

Exclusion Criteria:

* Unable to receive immunochemotherapy as first-line therapy due to co-morbidity or personal choice.
* Patients who have already started high dose steroids as a treatment for their lymphoma.
* Known diagnosis of infectious blood-borne virus e.g. Hep B, Hep C or HIV.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diffuse Large B Cell Lymphoma (DLBCL) or closely related high-grade B cell lymphomas including, but not limited to:
  * DLBCL NOS
  * Transformed follicular lymphoma
  * High grade B cell lymphoma with rearrangement of BCL2/BCL6 and MYC
  * Plasmablastic lymphoma
  * Primary Mediastinal Large Cell lymphoma
  * Burkitt lymphoma
  * Primary Central Nervous System lymphoma
  * High grade B cell lymphoma NOS
  Undergoing Standard of Care treatment for their lymphoma.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2020-09-17 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Establish a robust molecular monitoring pipeline. | 3-5 years
Successful identification of trackable mutations in collected samples. Feasibility will be met if more than 75% of the samples yield trackable mutations across the whole study. | 3-5 years

SECONDARY OUTCOMES:
Assess the utility of serial ctDNA assessment as a predicator of clinical outcome in high-grade B cell lymphoma. | 5 years
Assess the utility of integrated data from clinical risk factors (IPI), up-front genotype, serial ctDNA response and radiological assessment (CT or PET-CT). | 3-5 years
When the pipeline is optimised can these 4 parameters be available within 6 weeks, i.e. by completion of Cycle 2. | 3-5 years
  1. Clinical risk factors from the International Prognostic Index (IPI)
  2. Up-front genomic subtype based on molecular profiling of diagnostic biopsy
  3. Serial ctDNA monitoring during treatment.
  4. Radiological response imaging

OTHER OUTCOMES:
Identification of the de novo somatic variants in high-grade B cell lymphoma from collected ctDNA and tissue samples. | 3-5 years
Assess the utility of ctDNA to track clonal evolution in patients undergoing treatment for high-grade B cell lymphoma. | 3-5 years

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Hodson, PhD MRCP FRCPath, Principal Investigator — Cambridge University Hospitals NHS Foundation Trust
Locations (1):
- Cambridge University Hospitals NHS Foundation Trust, Cambridge, Cambridgeshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No